CLINICAL TRIAL: NCT01332799
Title: Xanthine Oxidase Inhibition in Renal Transplant Recipients
Acronym: XART
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Roberto S Kalil (Other)
Responsible Party: Sponsor-Investigator, Roberto S Kalil, Clinical Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201010787
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Complications of Renal Transplant
Keywords: cardiovascular disease; kidney transplantation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol (Active Comparator)
  Interventions: Drug: allopurinol or placebo
- Placebo (sugar pill) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: allopurinol or placebo — Daily active drug (allopurinol administered orally) administered orally for 3 years.
  Arms: Allopurinol
Other: Placebo — Sugar pill administered orally for 3 years.
  Arms: Placebo (sugar pill)

SUMMARY:
Cardiovascular disease is the leading cause of mortality in kidney transplantation. The enzyme xanthine oxidase may play an important role in the cardiovascular disease of kidney transplant recipients. Inhibiting this enzyme with allopurinol may improve vascular health and protects against cardiovascular complications.

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo controlled, clinical trial examining vascular effects of allopurinol in patients who received a kidney transplant that are maintaining stable renal function for at least 1 year. End-points include pulse-wave velocity, systemic blood pressure and kidney function among others.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* both genders
* recipients of living donor or deceased-donor kidney transplant with stable renal function

Exclusion Criteria:

* history of gout
* allergy to allopurinol
* use of azathioprine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto S Kalil, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Allopurinol: allopurinol Daily active drug (allopurinol administered orally)
- Placebo (Sugar Pill): Placebo: Daily placebo (sugar pill) administered orally for 3 years.
Period: Overall Study
Arm/Group | Allopurinol | Placebo (Sugar Pill)
Started | 10 | 10
Completed | 0 | 0
Not Completed | 10 | 10
Not completed — Insufficient funding | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Allopurinol; Placebo (Sugar Pill): allopurinol or placebo: Daily active drug (allopurinol administered orally) to be compared to daily placebo (sugar pill) administered orally for 3 years.
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Events
Description: Number of major cardiovascular events
Time Frame: 3 years
Population: No intervention occurred, so no data was collected for report.
Arm/Group | Allopurinol | Placebo (Sugar Pill)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Endothelial Function
Description: Changes in flow-mediated dilatation of braquial artery.
Time Frame: 3 years
Population: No intervention occurred, so no data was collected for report.
Arm/Group | Allopurinol | Placebo (Sugar Pill)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Arterial Stiffness
Description: Changes in pulse wave velocity.
Time Frame: 3 years
Population: No intervention occurred, so no data was collected for report.
Arm/Group | Allopurinol | Placebo (Sugar Pill)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study did not start
Description: Zero subjects considered 'at risk' for this study, as the intervention did not begin and zero subjects were at risk.
Arm/Group | Allopurinol | Placebo (Sugar Pill)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study did not receive funding so intervention did not begin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT01332799/Prot_SAP_000.pdf